CLINICAL TRIAL: NCT00812786
Title: Multicentre, Open Study for the Setting up of Population Pharmacokinetic Models and Bayesian Estimators for Individual Dose Adjustment of Immunosuppressive Drugs (Cyclosporine, Tacrolimus, Mycophenolate Mofetil, Everolimus) During the First Year Post-grafting in Adult Heart Transplant Recipients.
Brief Title: Pharmacokinetics of Immunosuppressive Drugs in Heart Transplant Patients
Acronym: PIGREC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006-006832-23
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2008-12

CONDITIONS: Heart Transplant
Keywords: heart transplantation; immunosuppressive drugs; individual dose adjustment; harmacokinetics; modelling
MeSH Terms: interventions — Cyclosporine; Tacrolimus; Mycophenolic Acid; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: cyclosporine, tacrolimus, mycophenolate mofetil and everolimus (immunosuppressive drugs)

SUMMARY:
The main objective is to develop pharmacokinetic methods for individual dose adjustment of the global immunosuppressive treatment (cyclosporine, tacrolimus, mycophenolate mofetil and everolimus, taking into account the pharmacokinetic interactions), in order to optimise the efficiency and reduce the potentially severe sides effects of these drugs.

Forty five heart-transplant patients are to be included in this phase IV study to obtain a minimum of 10 patients treated with tacrolimus-mycophenolate, 10 with cyclosporine-mycophenolate and 20 with everolimus-cyclosporine.

Ten to 11 blood samples will be collected within the 8 to 12 hours post-dose in each patient and the immunosuppressive drug concentrations will be measured by LC-MS/MS.

The pharmacokinetic models and Bayesian estimators thus developed will provide tools for individual dose adjustment of immunosuppressive drugs simultaneously, at different post-transplant periods, using the area under the concentration-time curve (AUC) estimated using a limited number of time-points (2 or 3).

DETAILED DESCRIPTION:
For each heart transplant patient, 10 to 11 blood samples (5 mL each) will be collected following dosing of he immunosuppressive drugs (at T0, T20', T40', T60', T90', T2h, T3h, T4h, T6h, T8h and T10h + T12h for inpatients), at several post-transplant periods (7 to 15 days, 1 month, 3 month and 1 year after transplantation). One more blood sample will be taken at D7-14 for pharmacogenetic analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patient having received of a heart transplant (exclusively) less than 2 weeks before the inclusion date or planned to receive it within days following inclusion.
* Patient at least 18 years old, male or female.
* Patient treated with one of the following combination : cyclosporine-mycophenolate, tacrolimus-mycophenolate or everolimus- "low-dose" cyclosporine for at least 3 days, and at least 24 hours by the oral route at the time of the first sampling day (between 7 and 15 days post-transplant).
* Patient included or not in another study, in particular in a therapeutic trial (e.g. comparison between drug combinations).
* Patient having given written informed consent for his/her participation to the trial.

Exclusion Criteria:

* Patients in disagreement with the present trial.
* Patients suffering from neuro-psychic problems, making them unable to well-understand the protocol or to give a reliable consent.
* Patients with previous heart or any other solid organ transplantation.
* Patients with double transplantation (heart-lung, heart-kidney or heart-liver)
* Patients still intubated and ventilated 15 days post-transplant.
* Patients with anaemia between Day 7 and 15, as characterized by hematocrit < 30% or haemoglobin < 9 g/dl.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-07; Primary Completion 2011-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Estimation of the pharmacokinetic properties and parameters of the immunosuppressive drugs.

SECONDARY OUTCOMES:
Investigation of relationships between physiological and pathological characteristics and individual pharmacokinetic parameters.
Characterisation of the exposure-clinical effects relationships for the difference immunosuppressive drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre MARQUET, MD, Principal Investigator — University Hospital, Limoges
Locations (12):
- France (12):
  - CHU de Bordeaux, Bordeaux
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Lille, Lille
  - CHU de Limoges, Limoges
  - Hôpital Louis Pradel - CHU de Lyon, Lyon
  - CHU de Nantes, Nantes
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CHU de Strasbourg, Strasbourg
  - CHU de NANCY, Vandœuvre-lès-Nancy

REFERENCES:
- [Result] Woillard JB, Saint-Marcoux F, Monchaud C, Youdarene R, Pouche L, Marquet P. Mycophenolic mofetil optimized pharmacokinetic modelling, and exposure-effect associations in adult heart transplant recipients. Pharmacol Res. 2015 Sep;99:308-15. doi: 10.1016/j.phrs.2015.07.012. Epub 2015 Jul 17. PMID 26192348